CLINICAL TRIAL: NCT03859310
Title: Precision of OCT and OCTA-based Ocular Measurements
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-53770
Record Dates: First submitted 2019-02-22; First posted 2019-03-01 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Normal Eyes and Ocular Pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Normal: no glaucoma or retinal pathology or corneal conditions
  Interventions: Device: SD-OCT
- Glaucoma: diagnosis of glaucoma
  Interventions: Device: SD-OCT
- Retina: diagnosis of AMD, DR or other retinal pathology
  Interventions: Device: SD-OCT
- Cornea: wear contact lens or prior refractive surgery or having dry eye or KCN
  Interventions: Device: SD-OCT

INTERVENTIONS:
Device: SD-OCT — Spectral Domain Optical Coherence Tomography for non-invasive, light-based, cross-sectional imaging of ocular structures

SUMMARY:
Precision of OCT- and OCTA-based Ocular Measurements

DETAILED DESCRIPTION:
The purpose of this study is to assess precision of measurements of vascular structures and the anatomical structures of the posterior pole of the eye based on OCTA and OCT scans in normal subjects, glaucoma patients, and retina patients, and to assess measurements of corneal layers based on corneal OCT scans in normal subjects and cornea patients.

ELIGIBILITY:
Inclusion Criteria:

* Normal - No glaucoma or treatment to lower IOP or retinal pathology for posterior imaging; No contact lens wear, dry eye, anterior pathology or ocular surgery for corneal imaging.
* Glaucoma - Have glaucoma and no history of other retinal pathology.
* Retina - Have retinal pathology and no history of glaucoma or treatment to lower IOP.
* Cornea - Contact lens wear or corneal condition such as dry eye, KCN, or post refractive surgery.

Exclusion Criteria:

* Normal - Unable to complete required exams; Clinical finding of posterior pathology or VA worse than 20/40 for posterior imaging; Clinical findings of corneal condition for corneal imaging.
* Glaucoma - Unable to complete required exams; Clinical signs of retinal pathology.
* Retina - Unable to complete required exams.
* Cornea - Unable to complete required exams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seeing eye doctor for routine care
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Repeatability and Reproducibility Standard Deviation of ocular measurements | Day 1
  calculated value minus the measured value

SECONDARY OUTCOMES:
Repeatability and Reproducibility Coefficient of Variation of ocular measurements | Day 1
  maximum difference that is likely to occur between repeated measurements

CONTACTS AND LOCATIONS:
Locations (1):
- AMA, Marysville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No